CLINICAL TRIAL: NCT02588040
Title: Post-Market Data Collection for Chronic Lateral Epicondylitis Patients Treated With Leukocyte- and Platelet-Rich Plasma (L-PRP) Prepared With the Recover Mini Platelet Separation Kit
Brief Title: Recover L-PRP in Lateral Epicondylitis (REGP-11-00)
Status: Terminated | Type: Observational
Why Stopped: Not enough sites available to complete enrollment in a timely manner
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BBIO.CR.LPRP.PMD.001.15
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Lateral Epicondylitis
Keywords: Chronic Lateral Epicondylitis; Leukocyte- and Platelet-Rich Plasma; Recover-L-PRP
MeSH Terms: conditions — Tennis Elbow | interventions — Leukocyte Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Leukocyte- and Platelet-Rich Plasma (L-PRP) — The Recover L-PRP Mini Platelet Separation Kit aids in the separation of the patient's own blood components by density through the use of a Biomet Biologics centrifuge.

SUMMARY:
The objective of the study is to further characterize the performance of L-PRP prepared using the Biomet Recover Kit in the treatment of chronic LE. The study will explore the potential impact of patient demographics and baseline characteristics on treatment outcome. Furthermore it will track and document treatment effects, time course, and untoward effects following treatment of chronic LE with L-PRP from the Recover device. In addition, the utilization of healthcare resources and associated costs will be investigated in treated patients.

DETAILED DESCRIPTION:
Clinical trials have been conducted to determine the efficacy and safety of Leukocyte- and Platelet-Rich Plasma (L-PRP) prepared with Biomet Recover L-PRP Mini Platelet Separation Kit for the treatment of tendinosis in a controlled setting. This study will allow for the capture and evaluation of real-world clinical data on a chronic LE patient population. The advantage of a post-market data collection is that it provides a way to examine clinical and patient reported outcomes along with the associated costs of chronic LE treatment in a diverse, clinically-relevant population. Although several registries exist which capture the outcomes following tendon/ligament reconstruction surgery, there are no known registries that capture outcomes following non-surgical treatment of chronic LE with Recover L-PRP. This study will fill that gap by allowing for an efficient data collection platform in a larger heterogeneous population of patients suffering from chronic LE and will document and more closely examine the treatment effects of Recover L-PRP.

ELIGIBILITY:
Inclusion Criteria:

1. Signed an independent ethics committee (IEC)-approved informed consent form (ICF).
2. Male or female of ≥ 18 years of age
3. Confirmed diagnosis of unilateral chronic LE
4. Duration of chronic LE symptoms ≥ 3 months
5. Failed at least one previous LE treatment (e.g. wait and see, physiotherapy, analgesics, NSAIDs, anti-inflammatory steroid injection and bracing, etc.).

   Exclusion Criteria:
6. No active systemic inflammatory condition (e.g., rheumatoid arthritis)
7. No active leukemia or metastatic malignant cells
8. No current chemotherapy treatments
9. No pregnancy
10. No lactation
11. No infected tendons, skin infection or skin disease in the area of the injection site.
12. Participating in another drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with chronic lateral epicondylitis (duration of symptoms ≥ 3 months)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study will be to measure number of patients who achieve resolution of chronic LE symptoms at 6 months following initial injection with Recover L-PRP. | 6 months

SECONDARY OUTCOMES:
Adverse events of interest | Evaluated at 3, 6, 12, 24 and 36 months
Numeric Rating Scale (NRS) | Evaluated at 3, 6, 12, 24 and 36 months
  Measure change in pain
Disability of the arm, shoulder and hand (QuickDASH) questionnaire | Evaluated at 3, 6, 12, 24 and 36 months
  Measure change in arm function
European Quality of Life 5 Dimensions 3 Levels (EQ-5D-3L) | Evaluated at 3, 6, 12, 24 and 36 months
  Measure change in quality of life
Resource utilization | Evaluated at 3, 6, 12, 24 and 36 months
  Cost of healthcare associated with chronic LE treatment
Number of injections of Recover L-PRP per patient in patients reaching symptom relief | Evaluated at 3, 6, 12, 24 and 36 months
Number of patients who have no recurrence of chronic LE within 36 months of the initial L-PRP injection | Evaluated at 3, 6, 12, 24 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Watts, MD, Principal Investigator — Wrightington Hospital, Wigan, United Kingdom
Locations (1):
- Wrightington Hospital, Appley Bridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided